CLINICAL TRIAL: NCT05199480
Title: Understanding the Impact of Cartridge-Based Electronic Cigarettes and Generated Aerosols on Cardiopulmonary Health
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: HM20022776
Record Dates: First submitted 2021-12-16; First posted 2022-01-20 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: E-Cig Use
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- E-cigarette liquid type 1 (Experimental): Participants will be instructed to use at least one study product daily in place of their own e-cigarettes during the intervention period.
  Interventions: Drug: Tobacco flavored liquid type 1
- E-cigarettes liquid type 2 (Active Comparator): Participants will be instructed to use at least one study product daily in place of their own e-cigarettes during the intervention period.
  Interventions: Drug: Tobacco flavored liquid type 2
- No e-cigarettes (No Intervention): No e-cigarette use

INTERVENTIONS:
Drug: Tobacco flavored liquid type 1 — A commercially available cartridge-based device with tobacco flavored liquid.
  Arms: E-cigarette liquid type 1
Drug: Tobacco flavored liquid type 2 — A commercially available cartridge-based device with tobacco flavored liquid.
  Arms: E-cigarettes liquid type 2

SUMMARY:
Over the last decade, e-cigarettes have become increasingly popular, due to their promotion as a healthy alternative to traditional tobacco cigarettes. However, there are large discrepancies of knowledge in understanding how these e-cigarettes affect the user's health. The overall goal of this study is to evaluate the impact of e-cigarettes usage on user's cardiopulmonary health

ELIGIBILITY:
Inclusion Criteria:

E-Cigarette group:

* 21 years of age or older
* Used e-cigarettes (≥3 times/week for ≥3 months)

Non e-cigarette group

● 21 years of age or older

Exclusion Criteria:

* 20 years old and younger
* Use of cigarettes for 15 days or more in the past 60 days
* Use of other tobacco products (cigars, hookah, smokeless) weekly or more frequently in the past 60 days
* Use of marijuana or any illicit or prescription drugs for non-medical use weekly or more frequently in the past 60 days
* Known allergy to propylene glycol or vegetable glycerin
* Evidence of cardiovascular, pulmonary, renal, hepatic, metabolic, or cerebral diseases
* Disorder or use of medication that affects cardiopulmonary health
* Evidence of pregnancy or current nursing

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Change in Peak oxygen consumption (VO2 peak) | Change from baseline to 2 weeks
  Participants' peak oxygen consumption (VO2 peak) will be measured using a standardized exercise capacity test performed on a stationary bike.
Change in Expiratory Volume | Change from baseline to 2 weeks
  Participants expiratory volume will be measured through spirometry using a pulmonary function device.

SECONDARY OUTCOMES:
Change in Skeletal muscle O2 utilization | Change from baseline to 2 weeks
  Assessment of skeletal muscle oxygen utilization using near-infrared spectroscopy through the ratio of O2 delivery and O2 extraction
Change in Maximal microvascular dilation | Change from baseline to 2 weeks
  Participants' microvascular function (maximal dilation) will be measured using local thermal hyperemia.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Rodriguez Miguelez, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2024-05-03): https://cdn.clinicaltrials.gov/large-docs/80/NCT05199480/Prot_000.pdf